CLINICAL TRIAL: NCT05756686
Title: Quantifying the Influence of Yogic Breathwork on Sleep
Brief Title: Influence of Yogic Breathwork on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Selda Yildiz, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00025528; R00AT010158 (NIH)
Record Dates: First submitted 2023-02-20; First posted 2023-03-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Sleep
Keywords: Sleep; Yogic Breathwork; Digital Health Technology; Yoga; Yogic Breathing; Slow Breathing; Sleep Tracking; Remote Research Studies; Wearable Devices
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Breathing Group 1 (Experimental): Arm 1 will receive an 8-week remotely delivered intervention that consists of a set of breathing practices through 60-minute weekly virtual group sessions (1day/week) with a 20-minute daily home sessions (in between weekly sessions; 6 days/week).
  Interventions: Behavioral: Breathing Group 1
- Breathing Group 2 (Active Comparator): Arm 2 will receive an 8-week remotely delivered intervention that consists of slow breathing practices through 60-minute weekly virtual group sessions (1day/week) with a 20-minute daily home sessions (in between weekly sessions; 6 days/week).
  Interventions: Behavioral: Breathing Group 2

INTERVENTIONS:
Behavioral: Breathing Group 1 — The 8-week breathwork intervention incorporates a set of breathing practices under the guidance of a certified yoga teacher.
  Arms: Breathing Group 1
Behavioral: Breathing Group 2 — The 8-week breathwork intervention incorporates a set of slow breathing practices under the guidance of a certified yoga teacher.
  Arms: Breathing Group 2

SUMMARY:
The purpose of this research study is to determine the influence of a regular yogic breathing practice on sleep, and to find out primarily if a regular practice of 8-week yogic breathing would enhance sleep quality as well as if it would improve participant's quality of life, and reduce existing stress. Study participants will be randomized into two arms for different breathing practices.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of two remotely-delivered 8-week breathing interventions on long term sleep patterns.

The study protocol consists of healthy participants (randomized in two breathing groups) undergoing a remotely delivered 8-week intervention and a 12-week sleep tracking period (including 2 week before the intervention, 8 week during the intervention, and 2 week after the intervention). Several sleep metrics will be extracted to characterize long-term sleep patterns and degree of sleep improvement. Participants will also be asked to complete pre- and post-intervention questionnaires.

The two remotely delivered interventions will be guided by two separate certified experienced yoga teachers. Both interventions will include 60-minute weekly group virtual sessions (1day/week) with a 20-minute daily home sessions (in between weekly sessions; 6 days/week) using home-aid practice materials.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* able to provide their consent to be in the study
* available and able to participate in study activities
* who can lie in supine
* who have little to no prior/current regular practice of breath awareness and training
* compatible devices for physiological data trackers

Exclusion Criteria:

* Inability to provide informed consent
* history of neurological disorders, craniospinal disorders, spinal injury
* diagnosed/treated sleep disorders such as sleep apnea with the use of CPAP
* allergic or respiratory disorders
* major or uncontrolled psychiatric illness or trauma or major depression
* lung and heart problems
* any condition requiring the use of medication that acts on the brain like stimulants/sedatives
* current substance abuse issues
* pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency (SE) | 12 weeks (8-week interventions and 2 weeks pre- and post-intervention period).
  SE is a measure ranging from 0 to 100% indicating the percentage time spent asleep relative to total time in bed. SE will be extracted during a 12-week period to then compute changes in SE.
Wake after sleep onset (WASO) | 12 weeks (8-week interventions and 2 weeks pre- and post-intervention period).
  WASO is the percentage of time spent awake during the remainder of the sleep period, after the first sleep onset. WASO will be extracted during a 12-week period to then compute changes in WASO.

SECONDARY OUTCOMES:
Total sleep time (TST) | 12 weeks (8-week interventions and 2 weeks pre- and post-intervention period).
  TST is the total time spent asleep. TST will be extracted during a 12-week period to then compute changes in TST.
Sleep latency (SL) | 12 weeks (8-week interventions and 2 weeks pre- and post-intervention period).
  SL is defined by the number of minutes spent awake in bed, prior to first sleep onset. SL will be extracted during a 12-week period to then compute changes in SL.
Pittsburgh Sleep Quality Index (PSQI) | During 2 weeks pre-intervention and 2 weeks post-intervention period
  PSQI is a self-reported questionnaire that is used to assess sleep quality. PSQI scores range from 0 to 21, with higher scores indicating worse outcome.
36-Item Short Form Survey Instrument (SF-36) | During 2 weeks pre-intervention and 2 weeks post-intervention period
  SF-36 is a self-reported questionnaire that is used to assess overall health. SF-36 scores range from 0 to 100, with higher scores indicating better health status.
Perceived Stress Scale (PSS) | During 2 weeks pre-intervention and 2 weeks post-intervention period
  PSS is a self-reported questionnaire that is used to measure the perception of stress. PSS scores range from 10 to 40, with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Yildiz, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: Study Pre-Screener Survey — https://octri.ohsu.edu/redcap/surveys/?s=3WW7YLDRTJFJWHME